CLINICAL TRIAL: NCT05215392
Title: A Smartphone Application of "Family Connections" to Increase the Use of Skills and the Improving of Psychological Symptoms in Relatives of People With Borderline Personality Disorder: a Protocol Study for a Randomized Controlled Trial.
Brief Title: A Smartphone Application of "Family Connections" to Relatives of People With Borderline Personality Disorder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJaumeI22-1
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Relatives
Keywords: borderline personality disorder; family connections; relatives; dbt; smartphone app; technology
MeSH Terms: conditions — Borderline Personality Disorder; Maple syrup urine disease, type 2

STUDY DESIGN:
Intervention Model Description: Randomized, Efficacy Study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (Experimental): Family members in the experimental group of this study will receive an ecological momentary intervention (EMI) derived from an ecological momentary assessment (EMA) via the Family Connections smartphone app.
  Interventions: Behavioral: Family Connections program
- Treatment As Usual (Active Comparator): Family members in this condition will receive the manual of Family Connections which contains all the information on the program sessions conducted and the skills training strategies in writing.
  Interventions: Behavioral: Family Connections program

INTERVENTIONS:
Behavioral: Family Connections program — Family members in the experimental group of this study will receive an ecological momentary intervention (EMI) derived from an ecological momentary assessment (EMA) via the Family Connections smartphone app. Family members in this condition will receive the manual of Family Connections which contains all the information on the program sessions conducted and the skills training strategies in writing.

SUMMARY:
The aims of our study are the following: (a) testing the effectiveness of a combined intervention: "Family Connections" program with a smartphone app versus the same intervention supported by a paper-based manual, (b) studying the feasibility and acceptance of both conditions and (c) evaluating the perceptions and opinions of families about both interventions.

DETAILED DESCRIPTION:
Family members of patients with borderline personality disorder (BPD) often experience high levels of suffering, anxiety, stress, burden and helplessness. The treatment program with the most empirical support is "Family Connections". It is one of the first programs specifically designed to help relatives of patients with BPD. The program is an adaptation of multiple strategies of Dialectical Behavioral Therapy. The results of these studies and their subsequent replications showed an improvement in family attitudes and perceived burden. Two of the technologies with very promising developments are Ecological Momentary Assessment and Ecological Momentary Intervention, that can act on each other. A large number of smartphone apps for people with psychological problems focus on the provision of instructions, adaptive self-help strategies, alarms, electronic diaries or emotional state ratings. The Family Connections app proposed in this article consists of a smartphone app built using EMA and EMI technologies.The aims of our study are the following: (a) testing the effectiveness of a combined intervention: "Family Connections" program with a smartphone app versus the same intervention supported by a paper-based manual, (b) studying the feasibility and acceptance of both conditions and (c) evaluating the perceptions and opinions of families about both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Having a family member diagnosed with borderline personality disorder.
* Being 18 years of age or older.
* Knowing and understanding the Spanish language.
* Having a smartphone with Internet connection.
* Completing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Burden Assessment Scale (BAS; Horwitz & Reinhard, 1992) | Changes will be assessed from pre-treatment to immediately after the intervention (3 months)
  Burden Assessment Scale (BAS) consists of 19 items and it assess the caregivers' objective and subjective burden within the past six months. Items are rated on a 4-point Likert scale ranging from 1(nothing) to 4 (a lot), and higher values indicate stronger burden. Internal reliability of the scale ranged from .89 to .91 and it shows adequated validity (Reinhard, Gubman, Horwitz & Minsky, 1994).

SECONDARY OUTCOMES:
Depression, Anxiety and Stress (DASS-21; Lovibond & Lovibond, 1995) | Changes will be assessed from pre-treatment to immediately after the intervention (3 months)
  Depression, Anxiety and Stress Scale (DASS) have 42 items about negative emotional symptoms (Lovibond & Lovibond, 1995). Lovibond & Lovinbod (1995) proposed that a part of these subscales for can become part of a short version creating a new questionnaire of 21 items. Items are rated on a 4-point Likert scale ranging from 0 (It did not happen to me) to 3 (It happened to me a lot or most of the time), and higher scores indicate worse symptoms of depression, anxiety or stress. DASS-21 showed fantastic factor structures. Regarding to the internal consistency, Cronbach's alphas were excellent for the DASS-21 subscales: Depression (α = .94), Anxiety (α = .87) and Stress (α = .91) (Antony, Bieling, Cox, Enns & Swinson, 1998).
Family Empowerment (FES; Koren, DeChillo & Friesen, 1992) | Changes will be assessed from pre-treatment to immediately after the intervention (3 months)
  Family Empowerment Scale (FES) consists of 34 items divided in three subscales: family, service system, and involvement in community that is refered to three ways of empowerment, attitudes, knowledge, and behaviors (Koren, DeChillo & Friesen, 1992). Items are rated on a scale of 1 (completely false) to 5 (totally true), and higher scores indicate a greater sense of empowerment. The psychometric properties are the following: regarding to the internal consistency of FES subscores, the coefficients ranged from .87 to .88 and validity and reliability are adequated (Koren, DeChillo & Friesen, 1992).
Resilience (CD-RISC; Connor & Davidson, 2003) | Changes will be assessed from pre-treatment to immediately after the intervention (3 months)
  Connor-Davidson Resilience scale is a 25-item measure of resilience. Items are rated on a 5-point Likert scale ranging from 0 (absolutely not) to 4 (almost always) and the punctuation is based on how the participant has felt over the last month. Higher scores means greater resilience (Connor & Davidson, 2003). The CD-RISC authors reported acceptable test-retest reliability (r = 0.87) and strong internal consistency (α = .89) (Connor & Davidson, 2003).

OTHER OUTCOMES:
System Usability Scale (SUS; Brooke, 2013). | Changes will be assessed immediately after the intervention (3 months)
  It consists of 10 items measured with a Likert scale with five response options from Strongly agree to Strongly disagree. It is reliable (coefficient alpha of .91) and useful (Bangor, Kortum, & Miller, 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Fernández Felipe, PhD Student, Principal Investigator — Universitat Jaume I; Diana Castilla López, Dr, Principal Investigator — University of Valencia; Mariví Navarro Haro, Dr, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication
Access Criteria: The data will be available to anyone who wishes to access them

REFERENCES:
- [Result] Hoffman PD, Fruzzetti AE. Advances in interventions for families with a relative with a personality disorder diagnosis. Curr Psychiatry Rep. 2007 Feb;9(1):68-73. doi: 10.1007/s11920-007-0012-z. PMID 17257517
- [Result] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Result] Hoffman PD, Buteau E, Hooley JM, Fruzzetti AE, Bruce ML. Family members' knowledge about borderline personality disorder: correspondence with their levels of depression, burden, distress, and expressed emotion. Fam Process. 2003 Winter;42(4):469-78. doi: 10.1111/j.1545-5300.2003.00469.x. PMID 14979218
- [Result] Hoffman PD, Fruzzetti AE, Swenson CR. Dialectical behavior therapy--family skills training. Fam Process. 1999 Winter;38(4):399-414. doi: 10.1111/j.1545-5300.1999.00399.x. PMID 10668619
- [Result] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Result] Rajalin M, Wickholm-Pethrus L, Hursti T, Jokinen J. Dialectical behavior therapy-based skills training for family members of suicide attempters. Arch Suicide Res. 2009;13(3):257-63. doi: 10.1080/13811110903044401. PMID 19590999